CLINICAL TRIAL: NCT05765487
Title: Phase 1 Single-Dose Double-Blind Vehicle-Controlled 3-Way Crossover Study Using Thermography to Assess the Pharmacodynamics and Pharmacokinetics of L-Arginine and Sildenafil Contained in Sildenafil Cream 3.6% in Normal Healthy Premenopausal Women
Brief Title: Using Thermography to Assess the Affects of Sildenafil Cream, 3.6%
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daré Bioscience, Inc. (Industry)
Collaborators: Strategic Science & Technologies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SST-6006-015
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Sexual Arousal Disorder
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Sildenafil Cream, 3.6% (Active Comparator): Contains both Sildenafil and L-arginine
  Interventions: Drug: Sildenafil
- Placebo Cream (Placebo Comparator): Contains L-arginine, no Sildenafil
  Interventions: Drug: Placebo
- Vehicle Cream (Other): Contains no L-arginine, no Sildenafil
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Sildenafil — Sildenafil Cream, 3.6%
  Arms: Sildenafil Cream, 3.6%
Drug: Vehicle — No Active or experimental ingredients
  Arms: Vehicle Cream
Drug: Placebo — Cream with only L-arginine
  Arms: Placebo Cream

SUMMARY:
The goal of this clinical trial is to compare thermography images in normal healthy premenopausal women after the application of Sildenafil Cream, 3.6%, L-arginine cream, and placebo cream. Participants will be shown a series of explicit videos to elicit a change in genital temperature before and after application of cream.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be a premenopausal woman at least 18 years of age.
* Subject must be willing to avoid high protein meals and follow dietary guidance provided by the study site staff for the duration of the study.
* Women of childbearing potential must be using an acceptable form of birth control (i.e., intrauterine system [IUS], progestin and/or estrogen-containing hormonal contraceptives, contraceptive patch, contraceptive implant, contraceptive ring, or contraceptive injection) or the copper-containing intrauterine device (IUD) and must be on a stable dose or have had the insert/implant for at least 1 month without complication prior to Visit 1 and agree to continue to stay on their birth control for the duration of the study. Condoms (latex or polyisoprene only) are not considered an acceptable form of birth control but may be used to prevent exposure to sexually transmitted infections. An attempt will be made to enroll at least 30% of women who are using hormonal contraception and at least 30% who are not.
* Subject reports she has viewed heterosexual pornography prior to Visit 1 and is sexually aroused from watching heterosexual porn or sexually explicit videos depicting men and women engaging in sexual activity.
* Subject has a body mass index (BMI) < 38 kg/m². Subjects with a BMI >30 kg/m2will be visually evaluated to ensure that there will not be physical interference with viewing the areas of interest by the thermography camera. If the investigator deems that interference is likely due to BMI, the subject will be excluded.
* Subject has a normal electrocardiogram at Visit 1.
* Subject is capable of understanding and complying with the protocol and agrees to sign the informed consent document.
* Subject has been sexually active (in the past 4 weeks since Visit 1). Sexual activity can include caressing, foreplay, masturbation, and vaginal intercourse.
* Subject is fluent in the English language.
* Subject is willing to trim pubic hair (if necessary) to allow for accurate genital temperature readings and visualization of the genital regions of interest.
* Subject has had a Pap smear performed within three years prior to Visit 1 and can provide documentation indicating results that are either normal or atypical squamous cells of undetermined significance (ASCUS) but negative for Human Papilloma Virus (HPV) (based on current guidelines as published by the U.S. Prevention Services Task Force). If the subject cannot provide documentation, a Pap smear will be performed at Visit 1. Subjects with abnormal findings will be excluded from study participation and be referred for follow-up medical care as appropriate.
* Subject is in good health for age, as determined by physical and gynecological history and examination at Visit 1.
* Subject agrees to withhold from smoking tobacco products 24 hours prior to all visits.
* Subject agrees to use compatible condoms (latex or polyisoprene) if she chooses to engage in vaginal or anal intercourse with her partner and abstain from receptive oral sex throughout the Double-Blind Dosing Phase and for seven days following the completion of Visit 4 to avoid potential partner exposure to the IP and to help prevent the transmission of sexually transmitted infections. Condoms should be used concurrently with subject's acceptable contraceptive method.
* Subjects must agree to not use vaginal or vulvar lubricants, spermicides, creams or gels, contraceptive foams, or vaginal douche products from Visit 1 until after the follow-up safety call is completed 7±3 days after Visit 4.

Exclusion Criteria:

* Subject is nursing or pregnant (based on positive urine pregnancy test) or wishes to become pregnant during the study period.
* Subject has any disorder or a history of any disorder that may prevent the successful completion of the study in the opinion of the Investigator.
* Subject has used any topical hormone replacement therapy (HRT) applied locally to the genitals in within three months of Visit 1.
* Subject has a significant cardiovascular, hepatic, metabolic, renal, respiratory, gastrointestinal, endocrine, immunologic, dermatologic, hematologic, neurologic, genitourinary, or psychiatric disease or other unstable medical condition that would contraindicate administration of study medication, interfere with study evaluation, limit study participation, or confound the interpretation of study results in the opinion of the Investigator.
* Subjects with controlled, treated thyroid disease on a stable medication for the past 6 months will be considered eligible. Thyroid Stimulating Hormone (TSH) must be within normal range (confirmed by laboratory test).
* Subjects with controlled, treated hypertension on a stable dose of ACE Inhibitors or Angiotensin II Receptor Blockers for the past 6 months will be considered eligible.
* Subject had an active ulcer or clinically significant bleeding disorder.
* Subject is actively menstruating at Visit 1 or has reported abnormal spotting in the 3 months preceding Visit 1.
* Subject has a history of myocardial infarction, stroke, or life-threatening arrhythmia within 6 months prior to Visit 1; or any history of coronary disease-causing angina; or congestive heart failure requiring medical intervention.
* Subject has retinitis pigmentosa or sickle cell anemia or related anemias, even if the subject feels clinically well at the time of Visit 1. Subjects with retinitis pigmentosa will be identified by specifically asking whether they have the condition, if there are visual signs and symptoms of the condition (including questioning subjects as to whether they have difficulty seeing at night or in low light, and if they have any visual field deficits that indicate a loss of peripheral or central vision), or if there is a family history.
* Subject has a history of orthostatic hypotension or orthostatic hypotension which is present at Visit 1, defined as a drop in systolic blood pressure ≥ 20 mm Hg, a drop in diastolic blood pressure ≥ 10 mm Hg or experiencing lightheadedness or dizziness at 1 or 3 minutes after the change in position from supine to standing.
* Subject reports a history of sexual dysfunction (e.g., anorgasmia, vaginismus, hypoactive sexual desire disorder, arousal difficulties etc.).
* Patient has dyspareunia, vulvovaginal infection or inflammation, inflammatory disorders of the vulva or vagina, vestibulodynia, clitorodynia, Genitourinary Syndrome of Menopause (GSM) or vulvovaginal atrophy.
* Subject has insulin dependent type 1 or type 2 diabetes.
* Subjects who do not demonstrate a greater positive slope for genital temperature change over time during the Sexually Explicit Video Session as compared to the Neutral Video Session during the 'no-cream' familiarization session at Visit 1 will not be eligible to advance into the Double-Blind Dosing Phase of the study. Any positive slope (i.e., any genital temperature increase, slope>0) during the sexually explicit file viewed in Visit 1 is considered qualifying for subjects to proceed into the double-blind dosing phase.
* Patient has undergone major pelvic surgery or abdominal surgery that may have caused nerve damage, including, vulvectomy and vestibulectomy.; neurological impairment due to diabetes, stroke, pelvic nerve damage secondary to trauma, cancer treatments, myasthenia gravis, multiple sclerosis or spinal cord damage.
* With the exception of anxiety and depression, patient has any current and/or previously reported diagnoses of DSM-IV-TR axis I disorders (e.g., schizophrenia, bipolar disorder) including delirium, dementia and amnestic disorders.
* Patients diagnosed with anxiety or depression must be controlled, as determined by the Investigator, and if on a medication (i.e., SSRIs, SNRIs, buspirone, bupropion and benzodiazepines), on a stable dose for at least the past 6 months.
* Patients who have any history of antipsychotic therapy within the last year will be excluded unless given for diagnosis of anxiety and/or depression and on a stable dose for the past 6 months if taking currently.
* Subject has a history of cancer, other than basal cell carcinoma.
* Subject has any surgical or medical condition that may interfere with the absorption, distribution, metabolism, or excretion of the test article in the opinion of the Investigator.
* Subject has a history of drug abuse within 1 year prior to Visit 1.
* Subject has a history of alcoholism within 1 year prior to Visit 1, admitted alcohol abuse, average consumption of more than 1 standard unit of alcohol per day (a standard unit equals 12 ounces of beer, 1½ ounces of 80-proof alcohol, or 6 ounces of wine).
* Subject has a history of non-arteritic ischemic optic neuropathy (NAION).
* Subject has had treatment currently or within 1 month (28 days) prior to Visit 1 with any of the following:

  1. Dehydroepiandrosterone (DHEA), excluding intravaginal DHEA, testosterone and other androgens, tamoxifen, raloxifene, and other selective estrogen receptor modulators (SERMs)
  2. Any antihypertensive (excluding ACE Inhibitors or Angiotensin II Receptor Blockers), clonidine, alpha blockers or nitrate containing medications.
  3. Beta blockers or other drugs that affect the autonomic nervous system and/or cardiovascular system
  4. Any approved or experimental medications or treatments used to enhance the sexual response (e.g., oral sildenafil, L-arginine)
  5. Any drugs or supplements that may alter amino acid or vitamin status, such as drugs or supplements containing L-arginine or Citrulline.
* Subjects who are currently being treated daily with weak, moderate, and strong inhibitors and inducers of CYP3A4 and CYP2C9 enzymes (e.g., CYP3A4: ketoconazole, clarithromycin, verapamil, diltiazem, St. John's Wort / CYP2C9: fluconazole, oxandrolone, fluvastatin, and metronidazole), Seville oranges, or any prescription, over-the-counter (OTC) medications, or herbal products known to inhibit or induce the 2 enzymes listed above must agree to continue taking the supplement or medication at approximately the same time each day for the duration of the study period, assuming the Investigator or subject's provider deems appropriate. If the subject is using the supplement or medication PRN, that subject must wash out (i.e., 6 half-lives) for the duration of the study period (Visit 1 to Visit 3), assuming the Investigator or subject's provider deems appropriate. If the subject takes any prescription or OTC drugs at the direction of a health care provider that are inhibitors or inducers of CYP3A4 and CYP2C9, that provider should be consulted before medications are stopped for the purposes of study participation.
* Subject has positive findings from the urine drug screen (e.g., amphetamines, barbiturates, benzodiazepines, cocaine, methadone, and opiates).
* Subject has positive findings for sexually transmitted infection (gonorrhea, chlamydia, trichomoniasis), or human immunodeficiency virus (HIV) antibodies.
* Subject reports having an outbreak (blisters, warts or vesicles) due to any of the following sexually transmitted diseases: genital herpes or HPV at any time point in the past three months.
* Subject has participated in any clinical research study evaluating another investigational drug or therapy within 30 days before Visit 1 (or 6 half-lives of the investigational agent, whichever is longer).
* Subject has any abnormal findings on vulvar-vaginal examination performed during the physical and gynecological exams at Visit 1 (e.g., genital skin breaks, irritation, dermatoses, or lesions).
* Subject has a genital piercing(s) or plans to get a genital piercing(s) during the study period which could interfere with thermal camera data collection or study objectives, as determined by the Investigator.
* Subject has moderate to severe current vaginitis, a vaginal infection including bacterial vaginosis (BV) or a yeast infection. The diagnosis of yeast infections should be made by the Investigator based on the physical and gynecological exams; the objective is to exclude women that are symptomatic. If the woman is not complaining of symptoms but the Investigator observes discharge, then a vaginal wet mount test should also be performed to confirm a diagnosis of yeast and Amsel criterion for confirmation of BV infection.
* Subject has a pelvic or urinary tract infection.
* Subject self-reports a known hypersensitivity to any ingredients in the Investigational Product (IP).
* Subject reports an orthopedic condition (e.g., labral tear, hip osteoarthritis) that may interfere with study participation, in the opinion of the Investigator, with regard to the thermography procedure during Visits 1 through 4.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 13 (Actual)
Dates: Start 2023-05-13 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
Evaluate the difference in vulvar blood flow after the use of investigational products | 14 days
  To evaluate and compare the impact of 2 grams of Sildenafil Cream 3.6%, Placebo Cream and Vehicle Cream on vulvar blood flow, as assessed by thermography in normal healthy premenopausal women.

CONTACTS AND LOCATIONS:
Locations (1):
- Pharma Medica Research, Inc., Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided